CLINICAL TRIAL: NCT00439257
Title: Costs, Quality of Life and Functional Outcomes in Veterans Treated for Multiple Sclerosis With Beta-Interferon l-B (Betaseron)
Status: Completed | Type: Observational
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Other Study IDs: SDR 94-001
Record Dates: First submitted 2007-02-21; First posted 2007-02-23 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2007-02

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1

SUMMARY:
The treatment of multiple sclerosis was evolving in light of specific drug therapies to treat the disease, refinements and acceptance of imaging with MRI to diagnose and monitor the disease process, and progress in understanding the pathogenesis of the inflammatory demyelinating process. The result was to raise new issues in the treatment of the disease, which are then being addressed by studies, including when to initiate treatment and the treatment of partial responders to existing therapies. Paralleling strides in treatment, and of particular importance to the Veterans Administration, was the effectiveness of such therapies, both in terms of cost to the VA Health Care System and quality of life of veterans with multiple sclerosis. This study addressed these issues.

DETAILED DESCRIPTION:
Background:

The treatment of multiple sclerosis was evolving in light of specific drug therapies to treat the disease, refinements and acceptance of imaging with MRI to diagnose and monitor the disease process, and progress in understanding the pathogenesis of the inflammatory demyelinating process. The result was to raise new issues in the treatment of the disease, which are then being addressed by studies, including when to initiate treatment and the treatment of partial responders to existing therapies. Paralleling strides in treatment, and of particular importance to the Veterans Administration, was the effectiveness of such therapies, both in terms of cost to the VA Health Care System and quality of life of veterans with multiple sclerosis. This study addressed these issues.

Objectives:

To consider how then currently used drug therapies for MS in veterans, e.g., Interferon beta-1b, interferon beta-1a and glatiramer acetate impact health related quality of life (HRQoL), physical function and disability and use of health care resources within the VA. Comparisons with other groups of veterans with specific chronic medical conditions will be made in order to develop a model of health care utilization based on indices derived from disability and impairment evaluations and HRQoL instruments.

Methods:

One hundred and twenty four veterans with a clinically definite multiple sclerosis at more than 30 VAMCs participated in this observational, prospective study. Prior to starting interferon beta-1b [IFNB-1b: Betaseron (tm)], interferon beta-1a [IFNB-1a: Avonex (tm)] or glatiramer acetate [Copaxone (tm)] baseline assessments were obtained: disability and impairment using the Kurtzke Expanded Disability Status Scale (EDSS) and Functional Scales (FS), and health related quality of life (HRQoL) using a veterans-modified version of the Short Quality of Life scale (SF-36V). Follow-up evaluations were performed at three months and every six months thereafter for three years. Veterans were monitored in terms of changes in their condition, side effects from drugs, and changes in therapies. Health utilization data obtained includes clinic stops, inpatient hospitalizations, cost of medications and supplies, training, referrals for prosthetics, rehabilitative therapies and long term care.

Status:

Completed.

ELIGIBILITY:
Inclusion Criteria:

Veteran enrolled at participating hospitals who have MS and are receiving the drugs of interest.

Exclusion Criteria:

Non-veterans or veterans not meeting the inclusion criteria.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 124 (Estimated)
Dates: Study Completion 2000-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph B. Guarnaccia, MD, Principal Investigator — VA Connecticut Healthcare System West Haven Campus, West Haven, CT; Robert M. Baumhefner, MD, Principal Investigator — VA Greater Los Angeles Healthcare System, West Los Angeles, CA
Locations (1):
- VA Connecticut Healthcare System West Haven Campus, West Haven, CT, West Haven, Connecticut, United States